CLINICAL TRIAL: NCT07011719
Title: A Randomized, Double-Blind, Active-Control, Multicenter Phase 3 Trial of Casdatifan and Cabozantinib Versus Placebo and Cabozantinib in Patients With Advanced Clear Cell Renal Cell Carcinoma
Brief Title: Study of Casdatifan and Cabozantinib Versus Placebo and Cabozantinib in Patients With Advanced Clear Cell Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEAK-1; 2024-515023-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma
Keywords: Casdatifan; Metastatic Clear Cell Renal Cell Carcinoma; Advanced Clear Cell Renal Cell Carcinoma; Kidney Cancer; PEAK-1; AB521; ccRCC
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental Arm) (Experimental): Casdatifan and cabozantinib taken orally
  Interventions: Drug: Casdatifan; Drug: Cabozantinib
- Arm B (Comparator Arm) (Placebo Comparator): Placebo and cabozantinib taken orally
  Interventions: Drug: Cabozantinib; Drug: Placebo

INTERVENTIONS:
Drug: Casdatifan — Administered as specified in the treatment arm
  Other Names: AB521
  Arms: Arm A (Experimental Arm)
Drug: Cabozantinib — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Arm B (Comparator Arm)

SUMMARY:
The purpose of the study is to evaluate the progression-free survival (PFS) of casdatifan versus placebo when each is given in combination with cabozantinib in adult patients with confirmed advanced or metastatic clear cell Renal Cell Carcinoma who have experienced progression on or after prior anti-PD-1 or anti-PD-L1 immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable and measurable locally advanced or metastatic renal cell carcinoma with a primary clear cell component.
* A Karnofsky Performance Status (KPS) score ≥ 80%
* At least 1 target lesion measurable by computed tomography/magnetic resonance imaging per RECIST 1.1, not within a field of prior radiation therapy.
* Adequate organ and marrow function, ≤ 72 hours prior to randomization.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test.

Exclusion Criteria:

* Received prior treatment with a HIF-2α inhibitor or cabozantinib.
* Other prior malignancy active within the previous year except for locally curable cancers that have been apparently cured.
* Clinically significant toxicities related to any prior anticancer treatment, or toxicities Grade ≥ 3 per National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0) regardless of relatedness to prior anticancer therapies.
* Uncontrolled or poorly controlled hypertension, as defined by a sustained blood pressure > 140/90 mm Hg on more than three antihypertensives
* History of leptomeningeal disease or spinal cord compression.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as assessed by Blinded Independent Central Review (BICR) according to RECIST 1.1 | up to approximately 33 months

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 64 months
Objective Response Rate (ORR) as assessed by Blinded Independent Central Review (BICR) according to RECIST 1.1 | up to approximately 33 months
Duration of Response (DOR) as assessed by Blinded Independent Central Review (BICR) according to RECIST 1.1 | up to approximately 33 months
Disease Control Rate (DCR) by Blinded Independent Central Review (BICR) | up to approximately 33 months
The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (SAEs) | up to approximately 33 months
Time to first symptom deterioration in National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy-Kidney Symptom Index - Disease Related Symptoms (NFKSI-DRS) Items 1-9 sub-scale score. | up to approximately 33 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (17):
- United States (17):
  - City of Hope - Phoenix Cancer Center, Goodyear, Arizona
  - City Of Hope National Medical Center, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Yale University, New Haven, Connecticut
  - Piedmont Cancer Institute OneOncology, Atlanta, Georgia
  - City of Hope Cancer Center Atlanta, Newnan, Georgia
  - City of Hope - Chicago Cancer Center, Zion, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Norton Cancer Institute PARENT, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Compass Oncology, OR, Portland, Oregon
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Tech University Health Science Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy